CLINICAL TRIAL: NCT02363114
Title: DOC Utility: Simple Screening of Depression, Obstructive Sleep Apnea and Cognitive Impairment to Identify Stroke Clinic Patients at Risk of Adverse Outcomes
Brief Title: DOC Utility: Screening of Depression, Obstructive Sleep Apnea and Cognitive Impairment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr. Richard H. Swartz (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Richard H. Swartz, Principle Investigator, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Other Study IDs: 141-2014; 1012404 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Stroke; Transient Ischemic Attack; Depression; Obstructive Sleep Apnea; Cognitive Impairment
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Depression; Sleep Apnea, Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stroke Prevention Clinic Patients: All consecutive patients presenting to six high volume Regional Stroke Prevention Clinics.

SUMMARY:
The primary objective of this study is to determine whether baseline DOC screening can add to clinical and demographic data to predict the occurrence of a composite negative outcome (any of: recurrent stroke, myocardial infarction, death, or admission to a long-term care (LTC) / complex continuing care (CCC) facility) within one year of screening, in stroke prevention clinic patients.

DETAILED DESCRIPTION:
The DOC screen will be routinely applied to all patients presenting to three high volume Regional Stroke Prevention Clinics (combined first visits >2,800 patients per year). Data will be abstracted from the patient chart using methodologies developed and validated in the Registry of the Ontario Stroke Network. The investigators have REB approval to collect this data and to link with administrative datasets through the Institute for Clinical and Evaluative Sciences (ICES). The investigators will use regression models to determine whether DOC screen scores add to baseline clinical and demographic data to predict the main negative outcomes. The investigators hope to identify which patients presenting to TIA/stroke prevention clinics are at highest risk of adverse long-term events so focused interventions can be developed to improve survival, outcomes and function of stroke prevention clinic patients.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients referred to regional stroke prevention clinics.
* This includes those discharged from hospital with a diagnosis of stroke or TIA, as well as emergency department referrals.
* The DOC CRF will also be completed for patients who are unable to complete the screen due to severe aphasia, severe motor dysfunction and language barriers (those who are not fluent in English without translation available).

Exclusion Criteria:

* Patients whose reason for referral to the clinic is neither Stroke nor TIA, as well as those who have been admitted to LTC/CCC facilities at the time of clinic visit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients attending outpatient Stroke Prevention and TIA Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with any Adverse Event | 1 Year from Initial Screen Date
  A composite negative outcome will be created, defined as the occurrence of any recurrent stroke, myocardial infarction, death, or admission to a long-term care (LTC) / complex continuing care (CCC) facility within one year of screening.

SECONDARY OUTCOMES:
Number of Participants with recurrent stroke | 1 Year from Initial Screen Date
  The number of participants with the occurrence of recurrent stroke within one year of screening
Incidence of DOC co-morbidities | 1 Year from Initial Screen Date
  To describe the incidence of DOC co-morbidities and outcomes in clinical important sub-groups (e.g. stroke-in-the-young, women vs. men, stroke in the "oldest-old" patients, TIA vs. ischemic stroke
Number of Participants with myocardial infarction | 1 Year from Initial Screen Date
  The number of participants with the occurrence of myocardial infarction within one year of screening
Number of Participants who died | 1 Year from Initial Screen Date
  The number of participants who died within one year of screening
Number of Participants who have been admitted to a long-term care or complex continuing care facility | 1 Year from Initial Screen Date
  The number of participants who have been admitted to a long-term care or complex continuing care facility within one year of screening

CONTACTS AND LOCATIONS:
Overall Officials: Richard H Swartz, MD, PHD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada